CLINICAL TRIAL: NCT02724670
Title: Single-arm Phase II Study of MR(Magnetic Resonance Imaging)-Based Image-guided Radiotherapy for Prostate Cancer
Brief Title: Study of MR-based IGRT for Prostate Cancer
Acronym: M-basePro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Arndt-Christian Mueller, PD Dr. med., University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-base Pro 1.0
Record Dates: First submitted 2016-03-10; First posted 2016-03-31 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiation (Other): IGRT 5x 2Gy/week, total dose: 78 Gy
  Interventions: Radiation: IGRT

INTERVENTIONS:
Radiation: IGRT — MR-based IGRT

SUMMARY:
MR (Magnetic Resonance Imaging) - based IGRT (image-guided radiotherapy) for patients with prostate carcinoma.

DETAILED DESCRIPTION:
Single arm, phase II study, MR (Magnetic Resonance Imaging) - based IGRT (Image-guided radiotherapy) of prostate cancer.

Primary endpoint: Grade 2+ GI (gastrointestinal) and genitourinary (GU) toxicity after 2 years.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven prostate cancer
* indication for curative treatment
* ECOG performance scale 0-2
* Informed consent

Exclusion Criteria:

* contraindications for curative treatment
* age<18year
* previous pelvic radiotherapy or prostatic treatment like TURP (transurethral resection of prostate), HIFU (high intensity focused ultrasound)
* serious comorbidity leading to inability for IGRT (image-guided radiotherapy)
* contraindications for MRI (Magnetic Resonance Imaging)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-03; Primary Completion 2020-06 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
G2+gastrointestinal and genitourinary toxicity at 2 years | Total trial treatment duration: 4 years, Duration for individual patient:Study treatment 9 months, Follow-up: 2 years for primary endpoint
  Number of participants with G2+-treatment-related genitournary and gastrointestinal adverse events assessed by CTCAE v4.0 and RTOG at 2 years

SECONDARY OUTCOMES:
Long-term GU-GI toxicity | 10 years after treatment
  Measurement of treatment-related genitournary and gastrointestinal adverse events assessed by CTCAE v4.0 and RTOG at 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Arndt-Christian Müller, Dr., Principal Investigator — Department of Radiation Oncology, University of Tübingen
Locations (1):
- Müller Arndt-Christian, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided